CLINICAL TRIAL: NCT00000668
Title: A Phase I Pharmacokinetic and Tolerance Study of 28-Day Regimens of Oral Ganciclovir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 127; ICM 1505; FDA 37A; RS-21592; 11102 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Retinitis; AIDS-Related Opportunistic Infections; Ganciclovir; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Retinitis; AIDS-Related Opportunistic Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — Ganciclovir

INTERVENTIONS:
Drug: Ganciclovir

SUMMARY:
To determine the pharmacokinetics (blood levels) of three dose treatment plans of oral ganciclovir during a 28-day dosing period. Other purposes of the study are to determine in a population of HIV seropositive persons with cytomegalovirus (CMV) viremia, the safety, tolerance, and patient acceptability of oral ganciclovir given for 28 days, to collect preliminary laboratory evidence for antiviral activity and effectiveness of three dose regimens of oral ganciclovir based on blood and urine cultures of CMV, and to relate antiviral activity to dosage and to serum ganciclovir levels.

CMV retinitis is an important sight-threatening opportunistic infection which affects about 10 to 15 percent of people with AIDS. A previous study has shown that treatment with ganciclovir resulted in a significant delay in time to first retinitis progression compared to untreated controls. More studies are warranted to evaluate effects at different doses.

DETAILED DESCRIPTION:
CMV retinitis is an important sight-threatening opportunistic infection which affects about 10 to 15 percent of people with AIDS. A previous study has shown that treatment with ganciclovir resulted in a significant delay in time to first retinitis progression compared to untreated controls. More studies are warranted to evaluate effects at different doses.

In group A, 36 HIV seropositive patients with CMV viruria receive a single dose of intravenous ganciclovir followed by one of three oral dose regimens for 28 days. Twelve individuals are treated at each dose level. In group B, 12 patients with AIDS and CMV retinitis receive oral ganciclovir therapy. These 12 patients must have received an induction course of intravenous ganciclovir for 4 weeks prior to study entry and must have stable CMV retinitis. Measurements for both groups include pharmacokinetics, safety, and tolerance (history, physical examination, hematology, and serum chemistry), and CMV blood and urine cultures. In addition, there are weekly ophthalmologic evaluations for individuals in the group B study.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Topical acyclovir.

There are two groups of patients. Group A must have:

* Confirmation of HIV infection by HIV antibody testing, p24 antigen, or culture of HIV.
* A positive urine culture for cytomegalovirus (CMV) within 4 weeks of study entry.
* Not received prior ganciclovir therapy.

Group B must have:

* A diagnosis of AIDS by CDC criteria.
* CMV retinitis diagnosed on funduscopic evaluation by an ophthalmologist.
* Completed 4 weeks of intravenous ganciclovir with an improvement or stabilization of retinitis. The course of therapy should include a minimum of 24 days total of intravenous ganciclovir.
* Patients in both groups must understand the nature of the study, agree to the tests required in the protocol, and must understand and sign an informed consent form approved by the appropriate Institutional Review Board (IRB) and by Syntex.

Required:

Group B:

* 4 weeks of intravenous ganciclovir which should include a minimum of 24 days total of intravenous ganciclovir.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Macular involvement due to cytomegalovirus (CMV) retinitis in both eyes.
* Active CMV retinitis in which there is progression.
* Presence of diarrhea or other clinically significant or uncontrolled gastrointestinal disease including persistent nausea and/or abdominal pain. Diarrhea is defined as > 3 unformed stools/day.
* Dementia or decreased mentation or other encephalopathic signs and symptoms which would interfere with the ability of the patient to follow the protocol, to take assigned dose regimen reliably, and to keep a daily record on a calendar.
* Significant CMV disease of other organs, including CMV gastroenteritis or CMV pneumonia.

Concurrent Medication:

Excluded:

* Any investigational drug.
* Acyclovir not specifically allowed.
* Any other nucleoside analog.
* Zidovudine (AZT).
* Probenecid.
* Aspirin.

Patients with the following are excluded:

* Macular involvement due to cytomegalovirus (CMV) retinitis in both eyes.
* Active CMV retinitis in which there is progression.
* CMV end organ disease.
* Presence of diarrhea or other clinically significant or uncontrolled gastrointestinal disease including persistent nausea and/or abdominal pain. Diarrhea is defined as > 3 unformed stools/day.
* Dementia or decreased mentation or other encephalopathic signs and symptoms which would interfere with the ability of the patient to follow the protocol, to take assigned dose regimen reliably, and to keep a daily record on a calendar.
* Significant CMV disease of other organs, including CMV gastroenteritis or CMV pneumonia.

Prior Medication:

Excluded within 4 days of study entry:

* Antimetabolite.
* Interferon.
* Other nucleoside analog including zidovudine (AZT).

Excluded for Group A:

* Ganciclovir or other anti-cytomegalovirus therapy.

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48
Dates: Study Completion 1995-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California
  - Davies Med Ctr, San Francisco, California
  - Mount Zion Med Ctr, San Francisco, California
  - Cornell Univ Med Ctr, New York, New York

REFERENCES:
- [Background] Spector SA, et al. Pharmacokinetic, safety and antiviral profile of oral ganciclovir in HIV-infected persons (ACTG 127). Natl Conf Hum Retroviruses Relat Infect (1st). 1993 Dec 12-16:154
- [Background] Spector SA, Busch DF, Follansbee S, Squires K, Lalezari JP, Jacobson MA, Connor JD, Jung D, Shadman A, Mastre B, et al. Pharmacokinetic, safety, and antiviral profiles of oral ganciclovir in persons infected with human immunodeficiency virus: a phase I/II study. AIDS Clinical Trials Group, and Cytomegalovirus Cooperative Study Group. J Infect Dis. 1995 Jun;171(6):1431-7. doi: 10.1093/infdis/171.6.1431. PMID 7769276